CLINICAL TRIAL: NCT00125346
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase 3 Trial to Assess the Efficacy and Safety of Tobramycin Inhalation Powder (TIP) in Cystic Fibrosis (CF) Subjects
Brief Title: Tobramycin Inhalation Powder (TIP) in Cystic Fibrosis Subjects
Acronym: EVOLVE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: per Data Monitoring Committee recommendation
Sponsor: Novartis (Industry)
Responsible Party: external affairs, novartis
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CTBM100C2301
Record Dates: First submitted 2005-07-28; First posted 2005-08-01 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Cystic Fibrosis
Keywords: Tobramycin Inhalation Powder
MeSH Terms: conditions — Cystic Fibrosis

INTERVENTIONS:
Drug: Tobramycin Inhalation Powder

SUMMARY:
Lung infections are a chronic problem for patients with cystic fibrosis (CF). Some patients with CF may have a type of bacteria called Pseudomonas aeruginosa in their lungs that can cause infections or make their symptoms worse. Tobramycin inhalation solution (TOBI) is an approved antibiotic, which is inhaled directly into the lungs, and can be used to manage these infections. Tobramycin inhalation powder (TIP) is a new, experimental powder formulation of tobramycin that is inhaled directly into the lungs using a T-326 inhaler. The purpose of this research study is to determine if TIP is safe and effective when compared to placebo (a powder with no medicine) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cystic fibrosis patients with Pseudomonas aeruginosa infection.
* Male and female subjects between 6 and 21 years of age at the time of screening.
* FEV1 at screening must be between 25% and 80% of normal predicted values.

Exclusion Criteria:

* Known local or systemic hypersensitivity to aminoglycosides or inhaled antibiotics.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Actual)
Dates: Start 2005-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) measured at week 1 and week 5.

SECONDARY OUTCOMES:
Time until first antipseudomonal antibiotic (an antibiotic used to treat bacteria of a certain type [the genus pseudomonas]) is used
Relative changes in FEV1 % predicted for patients who received TIP starting at visit 1 and for patients who received placebo starting at week 9, compared to all subsequent visits.
Relative change in FEV1 % predicted for patients who received placebo from week 5 to week 13
Relative change in FEV1 % predicted for patients who received placebo (from the average of four assessments [weeks 1, 2, 5, and 9] to week 13)
Change from baseline in susceptibility of pseudomonas to the antibiotic during the study measured at weeks 5, 9, 13, 17, 21, and 25, and change from baseline in quantity of pseudomonas found in sputum during the study measured at weeks 5, 9, 13, 17, 21,

CONTACTS AND LOCATIONS:
Locations (41):
- United States (26):
  - For information on a site near you, call 1-800-244-7668 Option "2", Mobile, Alabama
  - For information on a site near you, call 1-800-244-7668 Option "2", Phoenix, Arizona
  - For information on a site near you, call 1-800-244-7668 Option "2", Fresno, California
  - For information on a site near you, call 1-800-244-7668 Option "2", Long Beach, California
  - For information on a site near you, call 1-800-244-7668 Option "2", Los Angeles, California
  - For information on a site near you, call 1-800-244-7668 Option "2", Oakland, California
  - For information on a site near you, call 1-800-244-7668 Option "2", Sacramento, California
  - For information on a site near you, call 1-800-244-7668 Option "2", Orlando, Florida
  - For information on a site near you, call 1-800-244-7668 Option "2", Pensacola, Florida
  - For information on a site near you, call 1-800-244-7668 Option "2", Atlanta, Georgia
  - For information on a site near you, call 1-800-244-7668 Option "2", Augusta, Georgia
  - For information on a site near you, call 1-800-244-7668 Option "2", Chicago, Illinois
  - For information on a site near you, call 1-800-244-7668 Option "2", Oak Lawn, Illinois
  - For information on a site near you, call 1-800-244-7668 Option "2", Ann Arbor, Michigan
  - For information on a site near you, call 1-800-244-7668 Option "2", New Hyde Park, New York
  - For information on a site near you, call 1-800-244-7668 Option "2", New York, New York
  - For information on a site near you, call 1-800-244-7668 Option "2", Valhalla, New York
  - For information on a site near you, call 1-800-244-7668 Option "2", Durham, North Carolina
  - For information on a site near you, call 1-800-244-7668 Option "2", Cleveland, Ohio
  - For information on a site near you, call 1-800-244-7668 Option "2", Columbus, Ohio
  - For information on a site near you, call 1-800-244-7668 Option "2", Oklahoma City, Oklahoma
  - For information on a site near you, call 1-800-244-7668 Option "2", Philadelphia, Pennsylvania
  - For information on a site near you, call 1-800-244-7668 Option "2", Charleston, South Carolina
  - For information on a site near you, call 1-800-244-7668 Option "2", Tyler, Texas
  - For information on a site near you, call 1-800-244-7668 Option "2", Salt Lake City, Utah
  - For information on a site near you, call 1-800-244-7668 Option "2", Morgantown, West Virginia
- Argentina (2):
  - For information on a site near you, call 1-800-244-7668 Option "2", Buenos Aires
  - For information on a site near you, call 1-800-244-7668 Option "2", Córdoba
- Brazil (3):
  - For information on a site near you, call 1-800-244-7668 Option "2", Curitiba, Paraná
  - For information on a site near you, call 1-800-244-7668 Option "2", Florianópolis, Santa Catarina
  - For information on a site near you, call 1-800-244-7668 Option "2", Campinas, São Paulo
- For information on a site near you, call 1-800-244-7668 Option "2", Varna, Bulgaria
- Canada (3):
  - For information on a site near you, call 1-800-244-7668 Option "2", Vancouver, British Columbia
  - For information on a site near you, call 1-800-244-7668 Option "2", Hamilton, Ontario
  - For information on a site near you, call 1-800-244-7668 Option "2", Sainte-Foy, Quebec
- Chile (2):
  - For information on a site near you, call 1-800-244-7668 Option "2", Santiago
  - For information on a site near you, call 1-800-244-7668 Option "2", Viña del Mar
- For information on a site near you, call 1-800-244-7668 Option "2", Vilnius, Lithuania
- Mexico (3):
  - For information on a site near you, call 1-800-244-7668 Option "2", Mexico City
  - For information on a site near you, call 1-800-244-7668 Option "2", Monterrey
  - For information on a site near you, call 1-800-244-7668 Option "2", Tijuana